CLINICAL TRIAL: NCT02437695
Title: Robot Assisted Radical Prostatecomy and Positional Injury; 8 Years Survey
Brief Title: Robot Assisted Radical Prostatecomy and Positional Injury
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Other Study IDs: GK3
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Nerve Injuries
Keywords: Robotic Surgical Procedures; Trendelenburg Position
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although a condition for surgery, robotic interventions applied with steep Trendelenburg-lithotomy (ST-L) position may cause positional injury and peripheral neuropathy if good position is not achieved on the operating table. This study will be a 7-year retrospective examination of postoperative positional injury (PPI) in patients undergoing robot-assisted radical prostatectomy (RARP) for prostate diagnosis.

DETAILED DESCRIPTION:
Patients who underwent RARP between 2008-2014 will be evaluate. Patients with known peripheral neuropathy, lumbar-cervical discopathy, or history of orthopaedic surgery or trauma will exclude. The demographic data of patients, ASA, Charlson Comorbidity Index (CMI), Body Mass Index (BMI), operating time (OT) and Trendelenburg time (TT) will obtain from patient records. Patients will be questioned as to whether or not PPI had developed, if so, in which extremity, in what form (sensory-motor), duration, whether or not a doctor had been consulted, if so, what treatment had been given and whether or not the PPI had continued.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot-assisted radical prostatectomy (RARP) for prostate diagnosis.

Exclusion Criteria:

* Patients with known peripheral neuropathy,
* Lumbar-cervical discopathy,
* History of orthopaedic surgery or
* Trauma were excluded

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing robot-assisted radical prostatectomy (RARP) for prostate diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
retrospective examination of postoperative positional injury (PPI) in patients undergoing robot-assisted radical prostatectomy (RARP) for prostate diagnosis | 7 years
  The ST-L position carries high risk in terms of PPI, especially when lengthy surgery is planned and the risk could be increased in patients with high BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, MD, Study Chair — Unraniye training and research hospital
Locations (1):
- Istanbul Umraniye Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Mills JT, Burris MB, Warburton DJ, Conaway MR, Schenkman NS, Krupski TL. Positioning injuries associated with robotic assisted urological surgery. J Urol. 2013 Aug;190(2):580-4. doi: 10.1016/j.juro.2013.02.3185. Epub 2013 Mar 1. PMID 23466240